CLINICAL TRIAL: NCT06263998
Title: A Randomized, Double-blind, Parallel, Placebo-Controlled, Single and Multiple Ascending Dose Phase 1 Clinical Study to Assess the Safety, and Local Tolerance, Pharmacokinetics After Application of NCP112 Eye Drop in Healthy Subjects
Brief Title: Clinical Study for the Evaluation of Safety and Tolerability of NCP112 Eye Drops
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUC1-394
Record Dates: First submitted 2024-01-26; First posted 2024-02-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Xerophthalmia
MeSH Terms: conditions — Xerophthalmia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Single Ascending dose NCP112 Dose A (Experimental): NCP112 is administered once at a specified time in Day 1
  Interventions: Drug: NCP112
- Single Ascending dose NCP112 Dose A, Placebo (Placebo Comparator): NCP112 Placebo is administered once at a specified time in Day 1
  Interventions: Drug: NCP112 Placebo
- Single Ascending dose NCP112 Dose B (Experimental): NCP112 is administered once at a specified time in Day 1
  Interventions: Drug: NCP112
- Single Ascending dose NCP112 Dose B, Placebo (Placebo Comparator): NCP112 Placebo is administered once at a specified time in Day 1
  Interventions: Drug: NCP112 Placebo
- Single Ascending dose NCP112 Dose C (Experimental): NCP112 is administered once at a specified time in Day 1
  Interventions: Drug: NCP112
- Single Ascending dose NCP112 Dose C, Placebo (Placebo Comparator): NCP112 Placebo is administered once at a specified time in Day 1
  Interventions: Drug: NCP112 Placebo
- Multiple Ascending dose NCP112 Dose A (Experimental): NCP112 is administered twice daily. [time frame: Day 1- Day 14]
  Interventions: Drug: NCP112
- Multiple Ascending dose NCP112 Dose A, Placebo (Placebo Comparator): NCP112 Placebo is administered twice daily. [time frame: Day 1- Day 14]
  Interventions: Drug: NCP112 Placebo
- Multiple Ascending dose NCP112 Dose B (Experimental): NCP112 is administered twice daily.[time frame: Day 1- Day 14]
  Interventions: Drug: NCP112
- Multiple Ascending dose NCP112 Dose B, Placebo (Placebo Comparator): NCP112 Placebo is administered twice daily. [time frame: Day 1- Day 14]
  Interventions: Drug: NCP112 Placebo
- Multiple Ascending dose NCP112 Dose C (Experimental): NCP112 is administered twice daily.[time frame: Day 1- Day 14]
  Interventions: Drug: NCP112
- Multiple Ascending dose NCP112 Dose C, Placebo (Placebo Comparator): NCP112 Placebo is administered twice daily. [time frame: Day 1- Day 14]
  Interventions: Drug: NCP112 Placebo

INTERVENTIONS:
Drug: NCP112 — NCP112 topical ophthalmic solution
  Arms: Multiple Ascending dose NCP112 Dose A; Multiple Ascending dose NCP112 Dose B; Multiple Ascending dose NCP112 Dose C; Single Ascending dose NCP112 Dose A; Single Ascending dose NCP112 Dose B; Single Ascending dose NCP112 Dose C
Drug: NCP112 Placebo — Placebo comparator
  Arms: Multiple Ascending dose NCP112 Dose A, Placebo; Multiple Ascending dose NCP112 Dose B, Placebo; Multiple Ascending dose NCP112 Dose C, Placebo; Single Ascending dose NCP112 Dose A, Placebo; Single Ascending dose NCP112 Dose B, Placebo; Single Ascending dose NCP112 Dose C, Placebo

SUMMARY:
The objective is to evaluate the safety, local tolerability, and pharmacokinetics of NCP112 eye drops through single and multiple dose-escalation ocular administrations in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects aged 19 to 50 years at the time of screening (Visit 1).
2. Subjects with a body weight of 50.0 kg or more, and a body mass index (BMI) between 18.0 kg/m² and 30.0 kg/m² at the time of screening (Visit 1).

   ※ Body Mass Index (BMI, kg/m²) = Weight (kg) / [Height (m)]²
3. Subjects who have received sufficient explanation about the clinical trial, fully understand it, and have voluntarily decided to participate and signed the written informed consent.
4. Subjects deemed suitable as participants for this clinical trial based on the investigators judgment after physical examination, clinical laboratory tests, and medical history obtained during screening (Visit 1).

Exclusion Criteria:

1. Subjects with clinically significant diseases or history of diseases related to the liver, kidneys, cardiovascular system, gastrointestinal system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system (such as epilepsy, mood disorders, obsessive-compulsive disorder), hematologic/oncologic system, or urinary system (chronic or recurrent urinary tract infections).
2. Subjects with hepatitis B or C.
3. Subjects meeting any of the following criteria based on ophthalmologic history or examination during screening (Visit 1):

   * Corrected visual acuity of 20/40 or less.
   * Intraocular pressure exceeding 21 mmHg in either eye.
   * History of lacrimal drainage system disease or abnormal tear drainage.
   * History or suspicion of conditions affecting visual organs such as keratitis, iritis, uveitis, retinitis, dry eye syndrome, strabismus, glaucoma, etc.
   * Experience of adverse effects from contact lens use, or contact lens use within one month prior to the anticipated first dose, or inability to abstain from contact lens use during the clinical trial.
   * Ophthalmologic surgery (intraocular surgery) or laser vision correction surgery (such as LASIK) within 12 months prior to the anticipated first dose.
   * Silicone punctal occlusion or punctal cauterization within 3 months prior to the anticipated first dose (collagen punctal occlusion within 1 month).
   * Any other abnormal findings from ophthalmologic examination.
4. Subjects with a history of hypersensitivity to the active ingredients or excipients of the investigational drug, or to drugs in the same class as the active ingredients.
5. Subjects who have taken any medications related to dry eye syndrome (e.g., artificial tears, anti-inflammatory agents like cyclosporine, hyaluronic acid preparations, tetracycline preparations) or drugs that could induce dry eye syndrome or affect the outcome of this clinical trial (e.g., oral contraceptives, antihistamines, sedatives, oral aspirin, corticosteroids) within one month prior to the anticipated first dose.
6. Subjects who have taken any prescription drugs, eye drops other than those for dry eye, oriental medicine, or any other health supplements, including liver function supplements or vitamins within 2 weeks of the expected first dosing date, or any over-the-counter drugs within 1 week (unless other conditions are deemed appropriate by the investigator).
7. Subjects who have taken drug metabolism inducers or inhibitors, such as barbiturates, within one month prior to the expected first dosing date
8. Subjects with a history of drug abuse or a positive result on a urine drug test at screening (Visit 1).
9. Subjects unable to restrict grapefruit or grapefruit-containing food consumption from 7 days prior to the anticipated first dose through the duration of the clinical trial.
10. Subjects with systolic blood pressure of 90 mmHg or less, or 140 mmHg or more, or diastolic blood pressure of 50 mmHg or less, or 90 mmHg or more after sitting for at least 3 minutes without sudden postural changes during screening (Visit 1).
11. Subjects with a history of alcohol abuse, or who have consumed alcohol regularly (more than 21 units/week, 1 unit = 10 g = 12.5 mL of pure alcohol) within one month prior to the anticipated first dose, or are unable to abstain from alcohol during the clinical trial.
12. Subjects who regularly consume caffeine (e.g., coffee or green tea more than 5 units/day) or are unable to abstain from caffeine-containing foods from 24 hours prior to hospitalization through the duration of the clinical trial.
13. Subjects who have regularly smoked (including e-cigarettes, more than 10 cigarettes/day) within one month prior to the anticipated first dose, or are unable to abstain from smoking during the clinical trial.
14. Subjects who test positive on a breath alcohol test at screening (Visit 1).
15. Subjects who have participated in another clinical trial and received an investigational drug within 6 months prior to the anticipated first dose.
16. Subjects who have donated whole blood within 2 months, or component blood within 1 month, or received a blood transfusion within 1 month prior to the anticipated first dose, or who plan to donate or receive blood during the clinical trial.
17. Subjects who have received a vaccine within 14 days prior to the anticipated first dose or are expected to receive a vaccine during the trial period.
18. Female participants who test positive on a pregnancy test (urine hCG) conducted before the start of investigational drug administration, are pregnant, or are breastfeeding, except for those who have undergone surgical sterilization (Bilateral tubal ligation, Bilateral oophorectomy, or Hysterectomy).
19. Subjects who, during the entire clinical trial period and for at least 90 days after the last dose of the investigational drug, cannot or do not agree to use medically acceptable double contraception methods, or whose partner cannot or does not agree to use medically acceptable contraception, or who do not agree to refrain from donating sperm during this period.

    ※ Medically acceptable contraception methods include:
    * Use of an intrauterine device (IUD) with a documented failure rate by the partner.
    * Double contraception (use of barrier methods by both male and female partners).
    * Surgical sterilization of the subject or partner (vasectomy, tubal ligation, hysterectomy).
20. Subjects deemed unsuitable for participation by the investigator for other reasons (e.g., non-compliance with instructions).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Eye irritation(Likert scale) | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Local safety assessment
Eye redness(Likert scale) | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Local safety assessment
Intraocular pressure | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Opthalmic examination
History taking | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Opthalmic examination
Corrected vision test | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Opthalmic examination
Adverse events | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Including subjective and objective symptoms
Vital signs | Single dose Day -1 ~ Day 4, Multiple dose Day -1 ~ Day 22
  Blood pressure

SECONDARY OUTCOMES:
Cmax | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
AUClast | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
Tmax | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
AUCinf | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
t1/2 | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
CL/F | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
Vz/F | Day 1~Day 4 (Blood sampling at specified times within the time frame)
  Single dose - Evaluation of pharmacokinetic profile
Cmax | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
AUCtau | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
Cmax,ss | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
AUCtau,ss | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
Tmax | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
Cmin,ss | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
t1/2,ss | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
CLss/F | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
Vz,ss/F | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
PTF | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
R | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile
Tmax,ss | Day 1~Day 22 (Blood sampling at specified times within the time frame)
  Multiple dose - Evaluation of pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: INJIN JANG, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehak-ro, Jongno-gu, South Korea